CLINICAL TRIAL: NCT01757912
Title: Effect of Body Position Changes on Endotracheal Tube Cuff Pressure in Ventilated Critically Ill Patients.
Acronym: CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: General Hospital Sint-Blasius Dendermonde (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2010/668
Record Dates: First submitted 2012-12-21; First posted 2012-12-31 (Estimated); Last update posted 2012-12-31 (Estimated); Status verified 2012-12

CONDITIONS: Mechanical Ventilation With Oral Intubation
Keywords: mechanical ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cuff pressure after positioning (Experimental): The patient will be positioned in 16 distinct body positions. Immediately after correct positioning, the cuff pressure is measured.
  Interventions: Procedure: cuff pressure

INTERVENTIONS:
Procedure: cuff pressure — The patient will be positioned in 16 distinct body positions, immediately after correct positioning, the cuff pressure is measured during an end-expiratory ventilator hold.

SUMMARY:
The endotracheal tube secures free airway in patients undergoing surgical procedures or mechanical ventilation. The extraluminal airway needs to be sealed by a cuff. The cuff needs to be adequately inflated with air. The cuff pressure should be between 20 and 30 cm H2O. A cuff pressure in excess of the target range is associated with a risk of tracheal injury, whereas a cuff pressure below the lower limit includes a risk of micro-aspiration of subglottic secretions, with risk of subsequent ventilator-associated pneumonia. It is unknown whether the cuff pressure changes following changes in body position of the patient. The objective of this study is to investigate to which extent - if any - cuff pressures change after body position changes of the patient.

ELIGIBILITY:
Inclusion criteria are age 18 - 70 years, oral intubation with a taperguard EVAC endotracheal tube (Covidien®), conventional mechanical ventilation, adequate sedation (Richmond Agitation-Sedation Scale -5) and analgesia (Behavior Pain Scale 3 to 4).

Exclusion criteria are factors with potential influence on the cuff pressure or factors that disturbed the safety or well-being of the patient: pregnancy, palliative care, difficult intubation, decreased mobility of the neck, history of neck surgery, temperature of <35°C or >37.5°C, morbid obesity (body mass index >35) and every potential contra-indication for position changes such as unstable spinal cord injury or hemodynamic and/or respiratory instability.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
absolute values of cuff pressure (in cm H20) an number of measurement outside target range. | During surgical procedure or mechanical ventilation.
  Cuff pressure measurement will be executed with a universal pressure monitor.The patient will be positioned in 16 distinct body positions, immediately after correct positioning, the cuff pressure is measured during an end-expiratory ventilator hold. Cuff pressure is evaluated in the following 16 body positions: anteflexion of the head, hyperextension of the head, left lateral flexion of the head, right lateral flexion of the head, left rotation of the head, right rotation of the head, semirecumbent position with a 45° head of bed elevation, recumbent position with 10° head of bed elevation, horizontal backrest, trendelenburg 10°, left lateral position over 30°, 45° and 90°, and right lateral position over 30°, 45° and 90°.

CONTACTS AND LOCATIONS:
Overall Officials: Stijn Blot, PhD, Prof, Principal Investigator — University Ghent
Locations (1):
- General Hospital Sint Blasius, Dendermonde, Belgium

REFERENCES:
- See also: Related Info — http://www.uzgent.be